CLINICAL TRIAL: NCT06862271
Title: Comparison of Postoperative Analgesia, Delirium, and Parental Satisfaction Between Caudal Block Combined With General Anesthesia and Penile Block and Intravenous Fentanyl in Pediatric Urogenital Surgeries
Brief Title: Comparison of Caudal Block Combined With General Anesthesia and Penile Block and Intravenous Fentanyl in Pediatric Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Miray Gözde Özdemir (Other Government)
Responsible Party: Sponsor-Investigator, Miray Gözde Özdemir, Specialist / Doctor, Ankara Etlik City Hospital
Organization: Ankara Etlik City Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 102
Record Dates: First submitted 2025-02-28; First posted 2025-03-06 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Caudal Block; Pediatric Urologic Surgeries; Fentanyl; Pediatric Delirium; Analgesia
Keywords: pediatric urologic surgeries; pediatric delirium; caudal block; penile block; FLACC Scale; PAED Scale
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 ( Caudal block group ) (Active Comparator): In the caudal block group, after the induction of caudal block with investigations, 0.2% bupivacaine will be applied to the epidural space in a volume of 0.8 mL/kg and a maximum of 20 mL will be injected into the epidural space and the surgical incision will be made at the 15th minute.
  Interventions: Procedure: Group 1 ( Caudal block group )
- Group 2 (Penile block and IV Fentanyl group) (Active Comparator): In the penile block and IV fentanyl group, 1 µg/kg fentanyl will be administered by the investigations and 5 minutes later, penile block will be performed using 0.25% bupivacaine at a dose of 0.2 mL/kg.
  Interventions: Procedure: Group 2 (Penile block and IV Fentanyl group)

INTERVENTIONS:
Procedure: Group 1 ( Caudal block group ) — In the caudal block group, after the induction of caudal block with investigations, 0.2% bupivacaine will be applied to the epidural space in a volume of 0.8 mL/kg and a maximum of 20 mL will be injected into the epidural space and the surgical incision will be made at the 15th minute. For participants after surgery, Pediatric Anesthesia Emergence Delirium (PAED), Face Leg Activity Cry Consolability (FLACC) scales will be recorded, and for parental satisfaction, the LIKERT scale will be used. In addition, the child's walking time, first urination time, and need for additional painkillers will be questioned and recorded.
  Arms: Group 1 ( Caudal block group )
Procedure: Group 2 (Penile block and IV Fentanyl group) — In the penile block and IV fentanyl group, 1 µg/kg fentanyl will be administered by the investigations and 5 minutes later, penile block will be performed using 0.25% bupivacaine at a dose of 0.2 mL/kg. For participants after surgery, Pediatric Anesthesia Emergence Delirium (PAED), Face Leg Activity Cry Consolability (FLACC) scales will be recorded, and for parental satisfaction, the LIKERT scale will be used. In addition, the child's walking time, first urination time, and need for additional painkillers will be questioned and recorded.
  Arms: Group 2 (Penile block and IV Fentanyl group)

SUMMARY:
Urogenital surgery is one of the most frequently performed surgical procedures in the pediatric patient population. There is no consensus on which analgesic method is most effective for pain control in these patients. In clinical practice, if there are no contraindications, caudal block or penile block combined with intravenous fentanyl can be preferred as an analgesic method.

In this study, the results of these two analgesia methods will be compared with the research.Randomly selected participants will be compared by looking at parameters such as postoperative questionnaire results, walking time and urination time.

ELIGIBILITY:
Inclusion Criteria:

* 4 months - 12 years old male patient
* Acceptance of participation in the study
* Patients Planned for Urogenital Surgery
* ASA I-II Patients

Exclusion Criteria:

* <4 months, >12 years male patient
* Female patient
* Not accepted to be included in the study
* ASA status III-IV
* History of bleeding disorder
* Spinal cord disease
* Obstructive sleep apnea
* Developmental delay
* Behavioral disorder
* Allergy to any drug in the protocol

Ages: 4 Months to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Pediatric Anesthesia Emergence Delirium (PAED) Scale | The first evaluation will be made after extubation, the second evaluation will be made at the 15th minute after surgery.
  The PAED scale will be used to assess post-anesthesia emergence agitation. This scale was defined in 2004 and is considered the standard for diagnosing emergence agitation.
  The scale, consisting of five statements (from "child makes eye contact" to "child cannot be comforted") is rated from 1 to 4, with a maximum score of 20.
  Patients are observed for each of the 5 symptoms of delirium. After an observation is completed, the clinician subjectively scores the severity of that delirium symptom using the Lickert scale ("not at all," "only a little," "quite a bit," "very much," and "extremely"). A total score of 10 or more may be consistent with delirium urgent.
  As the score increases, a score of ≥10 points indicates 64% sensitivity and 86% specificity for delirium, while a score of >12 points provides 100% sensitivity and 94.5% specificity for the diagnosis of emergency delirium (ED).

SECONDARY OUTCOMES:
Face Leg Activity Cry Consolability (FLACC) Scale | The first evaluation will be made after extubation, the second evaluation will be made at the 15th minute after surgery.
  The FLACC scale will be used to assess pain. Developed as a tool for evaluating postoperative pain in children, this scale is one of the most widely known and commonly recommended pain measurement scales.
  Each category in the "FLACC" (Face, Legs, Activity, Cry, Consolability) pain assessment scale is evaluated between 0-2, Total score varies between 0 and 10.
  A score of 0 indicates that the child is calm and relaxed, a score of 1-3 indicates that the child is mildly disturbed, a score of 4-6 indicates that the child is in moderate pain, a score of 7-10 indicates that the child is significantly disturbed, in pain, or both.
LİKERT Scale | 24th hour after surgery
  The LIKERT scale will be used to assess the satisfaction of the patient and his/her parents. The Likert scale is a one-dimensional scale used to collect the opinions of the participants. In our study, a 5-point Likert scale will be used. The patient will be visited after the surgery, and the satisfaction of the patient and his/her relatives in the postoperative period will be questioned. 1) Not at all satisfied 2) Somewhat satisfied 3) Moderate 4) Very satisfied, 5) Excellent
  When comparing the groups, it will be evaluated that a higher LIKERT score constitutes 'better satisfaction'.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Yenimahalle, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No